CLINICAL TRIAL: NCT02554994
Title: The Effect of Multifactorial Intervention on Frailty in Vulnerable Older Adults Living in Rural Communities: A Designed Delay Trial
Brief Title: Multifactorial Intervention on Frailty in Vulnerable Older Adults
Acronym: ASPRA-IS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: PyeongChang Health Center & County Hospital (Unknown)
Responsible Party: Principal Investigator, Eunju Lee, Associate Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2015-0706
Record Dates: First submitted 2015-09-17; First posted 2015-09-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Frailty
Keywords: ASPRA cohort; multifactorial intervention; Medicaid services; Geriatric disorder; Short Physical Performance Battery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): ASPRA (Aging Study of PyeongChang Rural Area) cohort is a population-based, prospective cohort study of older adults living in PyeongChang County of South Korea. This cohort study is supported by public health center, named PyeongChang Health Center and Country Hospital managed by government, to improve the quality of aged public health services.
  All participants will be recruited from ASPRA cohort. After 6 months of usual care period, eligible participants are screened by characteristics of ASPRA database, and are assigned to a multifactorial intervention arm.
  Interventions: Other: Multifactorial intervention; Other: Usual care
- usual care (Active Comparator): The other participants enrolled to ASPRA cohort are acted as a control arm. The usual care according to ASPRA protocol will be maintained.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Multifactorial intervention — There are six components of intervention in this study.
  * For all participants:
    1. Group exercise
    2. Nutritional supplement(commercial liquid formula will be provided every day).
  * For selected participants:
    1. Wellness visit in primary care setting, polypharmacy and multi-morbidity every month.
    2. At risk of depression(the people identified as high risk of depression would meet psychiatrist every month).
    3. Domestic safety(If there are possible hazards in participants' home, social worker provide amendments for getting rid of it).
  Arms: Intervention
Other: Usual care — Experienced nurses will visit all participants every month during 6 months of study period, and will conduct an interview and comprehensive geriatric assessments to collect information regarding physical, nutritional, mental, mood condition and health related quality of life.
  According to ASPRA cohort schedule, all participants will be assessed by the composite measurement method composed of K-FRAIL frailty scare, Mini-Nutritional Assessment Short Form(MNA-S), the Korean version of Mini-Mental State Examination(K-MMSE), Center for Epidemiological Studies depression(CES-D), EQ-5D 3 level version from EuroQol Research Foundation(EQ-5D 3 level), Short Physical Performance Battery(SPPB), and the Cardiovascular Health Study(CHS).

SUMMARY:
Frailty is a highly prevalent, progressive condition in older adults that is characterized by multisystem physiologic impairments and vulnerability to stressful events, leading to increased risk of geriatric conditions, disability, falls, hospitalization, and mortality. An effective public health intervention to improve frailty in a rural aging population with limited resources remains unknown. The purpose of our study is to evaluate the effectiveness of multidimensional public health intervention to reduce frailty and related geriatric conditions in older adults in rural communities. Our hypotheses are that a multidimensional intervention consisting of group exercise, nutritional support, depression management, polypharmacy, and home safety intervention over a 6-month period will improve frailty and selected geriatric conditions in older adults who are in low socioeconomic status or living alone in a rural community. Our primary outcome is short physical performance battery at 6 month. Secondary outcomes include frailty status, nutritional status, depression, falls, sarcopenia, and health care utilization. The investigators will conduct a designed delay trial by implementing our intervention in one town for the first 6 months (intervention group), while measuring the outcomes without any intervention in another town (serving as a control group); in the following 6 months, the investigators will implement the 6-month intervention in the control town. The findings from our study will inform us to find effective public health interventions to promote healthy aging in resource-limited, rural populations.

ELIGIBILITY:
Inclusion Criteria:

1. Currently living in the PyeongChang county, GangWon province, South Korea
2. Aged 65 years or older
3. Living alone or receiving Medical aid services
4. Sign informed consent

Exclusion Criteria:

1. Unable to walk 100 meters, with or without assistive devices
2. Institutionalized for the past 6 months
3. Known metastatic cancer, end-stage heart disease, end-stage renal disease
4. Moderate to severe cognitive impairment (MMSE ≤ 18)
5. Plan to move out of the current residence in the next 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 187 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Improve the score of Short Physical performance battery | Change in every 6 months from baseline to end of the study

SECONDARY OUTCOMES:
Improve frailty index score calculated from the Cardiovascular Health Study criteria | Change at 6 months from baseline
Frailty status by the K-FRAIL criteria | Change at 6 months from baseline
Nutritional status by Mini-Nutritional Assessment Short Form(MNA-SF) | Change at 6 months from baseline
Depressive symptoms by Center for Epidemiologic Studies Depression Scale(CES-D) | Change in every 6 months from baseline to end of the study
Occurrence of falls | Change at 6 months from baseline
Sarcopenia measured by the consensus report of the Asian Working Group | Change in every 6 months from baseline to end of the study
Health care utilization(emergency room visit and hospitalizations) | Change at 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eunju Lee, Principal Investigator — Division of Geriatric Medicine, Department of Internal Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (2):
- South Korea (2):
  - PyeongChang Health Center & County Hospital, Gangwon-Do
  - Asan Medical Center, Seoul